CLINICAL TRIAL: NCT04285502
Title: Comparison of Postoperative Drain Insertion Versus No Drain Insertion In Patients Undergone Total Laparoscopic Hysterectomy
Brief Title: Comparison of Postoperative Drain Insertion Versus No Drain Insertion In Total Laparoscopic Hysterectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zeynep Kamil Maternity and Pediatric Research and Training Hospital (Other)
Responsible Party: Principal Investigator, enis ozkaya, ASSOCIATED PROFESSOR, Zeynep Kamil Maternity and Pediatric Research and Training Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZEYNEPKAMILHOSPITAL
Record Dates: First submitted 2020-02-22; First posted 2020-02-26 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: TOTAL ABDOMINAL HYSTERECTOMY
Keywords: surgical drain; visual analog scale; hematocrit

STUDY DESIGN:
Intervention Model Description: PROSPECTIVE RANDOMISED CONTROLLED TRIAL
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONTROL GROUP (No Intervention): patients without a drain
- CASE GROUP (Experimental): Patients a drain inserted
  Interventions: Procedure: SURGICAL DRAIN

INTERVENTIONS:
Procedure: SURGICAL DRAIN — A surgical drain is a tube used to remove blood, abscess and any type of fluid at the site of the place it is inserted
  Arms: CASE GROUP

SUMMARY:
This prospective randomized controlled trial was planned to be conducted among total laparoscopic hysterectomies performed at Zeynep Kamil Maternity and Children's Diseases Training and Research Hospital during one year period. The effect of drain insertion during the surgery will be assessed by this clinical trial. Patients will be assigned into two groups as cases and controls. Patients who will a drain inserted will be considered as case group and patients without a drain will be considered as control group. Patients will be evaluated according to their post operative VAS scores, hematocrit levels, their drainage volume and manifestation of an infection after the surgery.

DETAILED DESCRIPTION:
This prospective randomized controlled trial was planned to be conducted from February 2020 to February 2021 and included total laparoscopic hysterectomies performed at Zeynep Kamil Maternity and Children's Diseases Training and Research Hospital during the study period.

Surgeries on patients with existing comorbidity, with underlying malignant conditions, patients diagnosed deeply infiltrative endometriosis during surgery and patients who undergo multiple surgeries will be excluded from the study.

Clinical and descriptive data will be collected from both paper and electronic records, including the pain of the patient, the need for analgesia at the 6th-12th and 24th hour during the post-operative period. Visual analog scale (VAS) will be used to track the pain progression of the patients. Intraabdominal bleeding will be determined by measuring the hematocrit levels and drainage volume at postoperative day 1. Patients will also be assessed according to manifesting an infection in both the short term and long term.

Patients who will a drain inserted will be considered as case group and patients without a drain will be considered as control group. Data will be analyzed using the Statistical Package for Social Sciences (SPSS). A Chi-squared test will be used to evaluate the significance of the associations between variables. Continuous variables will be displayed as means and standard deviations. A P value of ≤0.050 will be considered as significant.

This study obtained ethical approval from the Medical Research & Ethics Committee of Zeynep Kamil Maternity and Children's Diseases Training and Research Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Female
* age between 40-70
* undergoing surgery for a benign condition
* having an abdominal surgery for the first time

Exclusion Criteria:

* existing comorbidity
* with underlying malignant conditions
* patients diagnosed deeply infiltrative endometriosis during surgery
* patients who undergone multiple surgeries

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2020-11-01 (Estimated); Study Completion 2021-02-01 (Estimated)

PRIMARY OUTCOMES:
analgesia need at the post-operative period | post operative 6. hour
  patient need for analgesia during post operative first day
hematocrit levels | post operative first day
  patient hematocrit level at post operative day 1
drainage volume | post operative first day
  drainage volume at postoperative day
post operative infection | post operative first day and post operative 1. week
  manifesting an post operative infection in short term and long term
pain post operative 6.-12. and 24. hour | pain
  will be measured using VAS score

SECONDARY OUTCOMES:
analgesia need at the post-operative 6. hour | post-operative 6. hour
  patient need for analgesia
analgesia need at the post-operative 12. hour | post-operative 12. hour
  patient need for analgesia

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Zeynep Kamil Maternity and Children Training and Research Hospital, Istanbul
  - Zeynep Kamil, Istanbul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Weston M, Soyer P, Barral M, Dohan A, Pierre S, Rabei R, Garcia-Reyes K, Kohi MP. Role of Interventional Procedures in Obstetrics and Gynecology. Radiol Clin North Am. 2020 Mar;58(2):445-462. doi: 10.1016/j.rcl.2019.11.006. PMID 32044017
- See also: Post-Caesarean Drain Placement - Minor Procedure Leading to Major Complication — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5324450/
- See also: The effect of peritoneal gas drain on postoperative pain in benign gynecologic laparoscopic surgery: a double-blinded randomized controlled trial — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4986969/